CLINICAL TRIAL: NCT04565691
Title: Bacteremia From Periodontal Treatment to Elucidate the Underpinnings of Sepsis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Collaborators: Skane University Hospital (Other); Swedish Dental Service Organisation (Unknown)
Responsible Party: Principal Investigator, Daniel Joensson, Associate Professor, Malmö University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lund university
Record Dates: First submitted 2019-01-29; First posted 2020-09-25 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Bacteremia; Periodontal Diseases; Sepsis; Heart Diseases
Keywords: Bacteremia; Periodontal disease; Sepsis; Heart Disease
MeSH Terms: conditions — Bacteremia; Periodontal Diseases; Sepsis; Heart Diseases

STUDY DESIGN:
Intervention Model Description: We study the impact of bacteremia. The subjects will be their own controls at the different time-points.
Masking Description: No masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bacteremia inducing arm (Experimental): As mentioned the participants will be their own controls at the different time-points.
  Interventions: Procedure: Non-surgical periodontal treatment

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Non-surgical periodontal treatment that is accepted to cause bacteremia in about 40% of the cases.

SUMMARY:
Approximately 40,000 Swedes suffer from sepsiseach year, about 20% die. Biomarkers that are sensitive to current or previous bacteremia are needed in the treatment of sepsis. Bacteremia from periodontal treatment is predictive and occurs in 13-75%. Cardiovascular disease (CVD) is the number one cause of death in industrialized countries and the impact of bacteria and their products need to be elucidated.

The study's hypothesis is to utilize bacteremia from periodontal treatment to evaluate biological markers for current or previous bacteremia.

A. What are the long term clinical, and 'omics related CVD-phenotypical effects from treating periodontal disease compared to an untreated group? B. Can biomarkers be used for detecting a bacteremia or previous bacteremia? C. Are the effects from bacteremia on cardiovascular biomarkers related to the individual's antimicrobial peptide profile? D. Does the presence of bacterial proteases, such as gingipain, relate to having a bacteremia from periodontal treatment and the systemic response from a bacteremia?

Significance: The project has the potential to shorten the time to treat sepsis, which in turn shortens hospital stay and higher survival. The possible definition of protective AMP-profile could translate to future pharmacologic intervention and improve the treatment of sepsis as well as prophylactic treatment at dental treatments. An elucidation of the impact of bacteria and their products on CVD could lead to personalized medicine targeting anti-inflammation and anti-oxidative stress in subjects with periodontitis.

As of March 2024 78 subjects have been included and we anticipate to keep the time-line that we set up.

DETAILED DESCRIPTION:
Bacteremia from periodontal treatment to elucidate the underpinnings of sepsis

Hypothesis In the context of cardiovascular disease (CVD) and sepsis this study hypothesise that (1) periodontal disease causes a specific CVD phenotype that can, to some extent, be reversed by treating periodontal disease; (2) that non-surgical periodontal treatment can be used as a human bacteremia model for evaluating biomarkers that can be used in the sepsis clinic; (3) that endogenous antimicrobial peptide profile dictate the severity of a bacteremia; (4) that proteinases from the oral biofilm can impact the severity of a bacteremia induced by oral bacteria and their products.

Aims A. What are the long term clinical, and 'omics related CVD-phenotypical effects from treating periodontal disease compared to an untreated group? B. Can biomarkers be used for detecting a bacteremia or previous bacteremia? C. Are the effects from bacteremia on cardiovascular biomarkers related to the individual's antimicrobial peptide profile? D. Does the presence of bacterial proteases, such as gingipain, relate to having a bacteremia from periodontal treatment and the systemic response from a bacteremia?

Project description To answer the clinical problems from the dental chair and the sepsis intensity care unit the investigators have designed the Bacteremia Study. Aim 1 is an intervention study, while Aim 2 and 3 are investigating the pathophysiological underpinnings of the association. When studying the long term effects of periodontal treatment on CVD phenotype Malmö Offspring Dental Study (MODS) participants who have not sought dental care despite being told they have periodontal disease, will be invited as non-treated controls. The primary outcome variable will be changes in total carotid plaque area (TPA) per year.

In Aim 2 and 3 the parameters used to dissect the different aspects of the bacteremia. The AMP profile may be different in subjects with more severe bacteremia (measured by blood culturing) versus no bacteremia. The primary outcome will be concentration of CVD biomarkers during and following bacteremia (positive blood culture) compared to those who have negative blood culture.

Recruitment The participants are recruited at the Swedish Dental Service of Skåne in Lund, at the Department for Periodontics. The inclusion criteria is having periodontal disease - one quadrant with ≥2 teeth with > 5mm pocket depth (PD) and this quadrant will be treated when the blood samples are taken. The treatment is mechanical non-surgical periodontal treatment. Exclusion criteria is having a conditions that require prophylactic antibiotics at periodontal treatment.

Number of recruited participants The study will recruit 100 participants plus reexamination of MODS participants who have not sought periodontal treatment. Unfortunately, the available literature on bacteremia at periodontal treatment is very heterogeneous (13-75%), making it difficult to perform a meaningful power calculation. The investigators have decided on 100 participants and this has been approved by the Ethical Review Authority.

Cardiovascular phenotyping At baseline and after 1 year and 2 years the participants undergo cardiovascular phenotyping at Clinical Research Unit at Skåne University Hospital (Kliniska Forskningsenheten, KFE). The cardiovascular phenotyping in this project is based on several subclinical parameters mentioned bellow, however the most important is carotid artery ultrasound for assessment of carotid plaque area and stability. Associate Professor Jönsson is the first author and Olle Melander co-author of a publication investigating the association between periodontal disease and carotid total plaque area has. The carotid imaging in this project is performed by the same personal using the same equipment as in Jönsson et al..

• Carotid artery ultrasound (GE logiq E9) of both carotids.

* Presence of carotid plaque.
* Number of carotid plaques.
* Area of carotid plaque(s).
* Visual cap.
* Degree of stenosis.
* Gray scale medium (GSM) of carotid plaque.
* Statistical geometric feature (SGF) - spottiness of the plaque. The GSM and SGF (actually SGF/plaque area or SGF/degree of stenosis) is an expression of heterogeneity of the plaque on ultrasound and is correlated to plaque area stained for lipids, macrophages and hemorrhage as well as cytokine expression. While GSM gives the overall echogenicity in the plaque, SGF is a measurement that describe the distribution of grey scale levels within the plaque.

Other parameters in cardiovascular phenotyping included in the project:

* Blood pressure - sitting blood pressure.
* BMI and hip/waist measurement.
* Total cholesterol (TC), LDL-C and HDL-C.
* Fasting blood glucose (FBG) and HbA1c.
* GWAS for genes associated with CVD. Blood culture and blood 16S sequencing At all time-points blood is drawn for culturing and blood 16S-sequencing analysis. For culturing the phlebotomists in the study have been trained by the nurses at the infection clinic on how to draw blood for culturing - 4 blood culturing flasks per time point - one anaerobe and one aerobe on each arm.

Blood will be drawn and DNA will be extracted from PBMCs. For subsequent sequencing 16S amplicon sequencing will be used with amplicon sequencing variants (ASV) based bioinformatics pipeline, which increases the resolution and allows a larger fraction of the bacteria to be identified with species resolution. The results from the blood 16S sequencing will then be compared to the content of the oral biofilm.

Biomarkers The biomarkers play two important roles in this project - firstly, they are biomarkers of bacteremia that the investigators evaluate, and the sequencing of blood bacteria is also considered to be a biomarker of previous bacteremia, as described above. Secondly, and perhaps even more importantly, they collectively reflect the systemic response. Bacteremia can initiate sepsis, but the host response is what causes the condition.

For the analysis the biomarkers are divided into those immediately sent to the hospital lab, and biomarkers that the investigators analyze when all samples are collected. The biomarkers analyzed immediately are

* Procalcitonin (PCT)
* High sensitivity troponin T (hsTNT)
* High sensitivity C-reactive protein (hs-CRP)
* N-terminal prohormone of brain natriuretic peptide (NT-proBNP)

In a later phase, the investigators will also analyze:

* Mid-regional pro-adrenomedullin (MR-pro-ADM)
* C-terminal pro-endothelin-1 (CT-pro-ET-1)

When the investigators collected all samples, the investigators will utilize a multiplex approach for novel biomarker detection, such as OLINK proteomics.

Antimicrobial peptides Antimicrobial peptides will be analyzed by quantitative selected reaction monitoring mass spectrometry (SRM-MS), in accordance with previously published work from the group.

Proteases Proteases, and especially gingipain form Porphyromonas gingivalis has gained attention through a recent publication reporting on the effects from gingipain on the disease progression of Alzheimer's disease. Proteinases and gingipain specifically, will be analyzed in GCF, and also in plasma. Thanks to previous funding the investigators have, in collaboration with Innovagen, created anti-gingipain antibodies that will be evaluated.

Statistics Aim 1 statistics - The intervention trial aspect will be primarily based on changes in carotid total plaque area (TPA). The annual change in TPA will first be assessed in the non-treated subjects from MODS. Changes in TPA will be treated as a dependent variable in a linear regression. Periodontal treatment versus untreated control will be used as independent variable. Other independent variables will be confounding factors, such as age, smoking status, education, medication, blood pressure etc. The investigators will then continue by using 'omics related biomarkers, such as OLINK proteins, as independent variables.

Aim 2 statistics - To investigate the association between cardiovascular biomarkers and bacteremia the investigators will investigate each time-point (Figure 1) separately. To investigate the association between bacteremia and CVD biomarkers, positive blood culture / previous blood culture / colony forming units (CFU) will be used as dependent variables and the biomarkers as independent variables in logistic/linear regressions, adjusting for confounders. ROC-curves will be constructed to test biomarkers of bacteremia at the respective time-points, to predict positive blood culture / previous blood culture.

Aim 3 statistics - To assess the impact of the AMP-profile, individual peptides will be included in a principal component analysis (PCA). A linear regression model with biomarkers as dependent variables and blood culture and PCA factors as independent variables will be constructed.

Aim 4 statistics - Proteases will be included as independent variables in logistic and linear regression models with blood culture and biomarkers as dependent variables, respectively.

The results from sequencing blood for microbiome will be analyzed in relation to the effects on biomarkers and blood culture, respectively, in the aims of 3 and 4.

Significance A thorough investigation of the underpinning of the association between CVD and periodontal disease and how periodontal disease may impact the course of CVD will be important in understanding the association. Decades of frequent low grade bacteremia may have caused more severe damages to the cardiovascular system in need of more personalized attention from cardiologists. This study elucidates what that cardiologist should look for.

In the context of sepsis the current project has the potential to contribute to more sepsis patients surviving the disease through a more precise and faster targeting of the bacteria initiating the condition. A biomarker that is more sensitive to bacteremia than blood culture and allows fast analysis would contribute to shorter time to correct antibiotics, which is the most important factor for shorter hospital stay and less deaths from sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Periodontal disease

Exclusion Criteria:

* Recently used antibiotics.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Bacteremia | At baseline, periodontal treatment (within 5 min) and 1 hour, 1 day, 1 week and 1 year after periodontal treatment.
  Changes in positive blood culture

SECONDARY OUTCOMES:
Changes in levels of biomarkers in relation to bacteremia | At baseline, periodontal treatment (within 5 min) and 1 hour, 1 day, 1 week and 1 year after periodontal treatment.
  Changes in levels of biomarkers following bacteremia

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Jonsson, DDS PhD, Principal Investigator — Malmo University, Lund University
Locations (1):
- Folktandvarden Skane, Lund, Sweden